CLINICAL TRIAL: NCT05077371
Title: Peer Support Program in cáncer Patients Elkar Laguntza
Brief Title: Peer Support Program in Cancer Patients Elkar Laguntza
Acronym: ElkarLaguntz
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joana Perez Tejada (Other)
Collaborators: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Sponsor-Investigator, Joana Perez Tejada, Psychology researcher, Onkologikoa
Organization: Onkologikoa (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PI2018068; 2019 (Other: Kutxa Fundazioa)
Record Dates: First submitted 2021-09-21; First posted 2021-10-14 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Neoplasms; Social Skills; Psychological Distress
MeSH Terms: conditions — Neoplasms; Social Skills

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group 1 (Experimental): newly diagnosed breast cancer patients receiving the peer support program at the beginning of their medical treatment.
  Interventions: Behavioral: Peer support program
- Experimental group 2 (Experimental): newly diagnosed breast cancer patients receiving the social peer support program at the end of their medical treatment.
  Interventions: Behavioral: Peer support program

INTERVENTIONS:
Behavioral: Peer support program — The intervention will consist of 8 face-to-face peer social support sessions conducted by volunteers diagnosed with breast cancer who have finished their medical treatment (chemotherapy, radiotherapy, surgery) or who have been in a stable phase for at least two years and who are motivated to participate in this type of intervention.

SUMMARY:
In cancer patients, social support provided by partners, family and/or friends plays a key role in coping with the disease and reducing treatment-related distress. However, research indicates that some of the needs of patients, such as coping with the disease, reducing isolation or managing guilt, often go unmet. With the aim of trying to meet these types of needs of people with cancer, the present research will evaluate the effectiveness of a peer support program in cancer patients, based on the support provided or exchanged by people who have faced similar challenges or problems. The intervention will consist of 8 face-to-face sessions of social peer support, involving a cancer patient and a volunteer who is in a stable phase and who has undergone the same diagnosis and medical treatment. To evaluate the effectiveness of the social support program, the immediate and long-term effect of participation in the program on both psychological (anxious-depressive symptoms, quality of life, perception of the disease, coping strategies, perception of social support,...) and biological (endocrine and immune system) variables will be analyzed.

DETAILED DESCRIPTION:
The general aim of the present research will be to evaluate the effectiveness of a peer social support intervention in cancer patients at the Onkologikoa Foundation of Guipuzcoa. Specifically, the immediate and long-term effect that such intervention will have on symptoms of psychological distress, quality of life, coping strategy, perception of social support, perception of the disease and emotional regulation will be evaluated. As a secondary aim of this study, we intend to evaluate the immediate and long-term effect of the peer social support intervention on the immune system (through the determination of the levels of cytokines IL-1β, IL-2, IL-6, IL-8, IL-10, IFN-γ and TNF-α), on the monoaminergic system (through the determination of plasma levels of serotonin, tyrosine, phenylalanine, tryptophan, quinurenine, quinurenic acid and 3-HK), on the HPA axis (through the measurement of the diurnal cycle of cortisol), and on sex hormones (through the measurement of estradiol and testosterone levels), systems that have been related both to the development of anxious-depressive symptoms and to the development, progression and recurrence of cancer.

In addition, it will be studied at what time the application of the program is most effective, being applied in newly diagnosed patients (experimental group 1) and in patients who have just finished medical treatment (experimental group 2).

ELIGIBILITY:
Inclusion Criteria:

* having received the diagnosis of cancer in the last month; not having started medical treatment; the tumor type and medical treatment coinciding with any of the volunteers.

Exclusion Criteria:

* relapse; suffering or having suffered from a severe mental disorder (according to DSM-V criteria).

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychological distress scale HADS | baseline
  Hospital Anxiety and Depression Scale ( HADS) was originally developed by Zigmond and Snaith (1983) and is commonly used by doctors to determine the levels of anxiety and depression that a person is experiencing. The total score is out of 42, (21 per anxiety and 21 per depression). Higher scores indicate greater levels of anxiety or depression.
Social support perception scale MOS-SSS | baseline
  The Social Support Scale (MOS-SSS) aims to assess the extent to which the person has the support of others to face stressful situations. 19 items with answer categories that range on a 7-point rating scale. Higher scores indicate greater levels of social support perception
Coping scale COPE28 | baseline
  The COPE inventory was created by Carver (1989). It is a multi-dimensional inventory developed to asses the different coping strategies people use in response to stress. Self-distraction, items 1 and 19 Active coping, items 2 and 7 Denial, items 3 and 8 Substance use, items 4 and 11 Use of emotional support, items 5 and 15 Use of instrumental support, items 10 and 23 Behavioral disengagement, items 6 and 16 Venting, items 9 and 21 Positive reframing, items 12 and 17 Planning, items 14 and 25 Humor, items 18 and 28 Acceptance, items 20 and 24 Religion, items 22 and 27 Self-blame, items 13 and 26. Range: 2-8. Higher scores indicate greater levels of coping
Resilience scale | baseline
  The Resilience Scale (RS) was developed to evaluate the levels of resilience in the general population. The items are rated on a 7-point scale ranging 1 (strongly disagree) to 7 (strongly agree), with a score ranging 14 to 98. Higher scores indicate greater levels of resilience
Quality of life scale SF-12 | baseline
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It consists of physical and mental component scores (PCS/MCS), ranging from 0 to 100. Higher scores indicate greater quality of life.
emotional inteligence scale TMMS | baseline
  The Trait Meta-Mood Scale (TMMS; Salovey, Mayer, Goldman, Turvey, & Palfai, 1995) is a well-established measure of perceived emotional intelligence, an aspect of emotional intelligence that includes people's beliefs and attitudes about their own emotional experience. The TMMS-24 contains three key dimensions of emotional intelligence with 8 items each: Emotional Attention, Emotional Clarity and Emotional Repair. The score ranges from 7 to 56. Higher values indicate higher emotional intelligence
illness perception scale | baseline
  The Illness Perception Questionnaire (IPQ) is a widely used multifactorial pencil-and-paper questionnaire which assesses the five cognitive and emotional illness representations and comprehensibility. Five of the items assess cognitive illness representations: consequences (Item 1), timeline (Item 2), personal control (Item 3), treatment control (Item 4), and identity (Item 5). Two of the items assess emotional representations: concern (Item 6) and emotions (Item 8). One item assesses illness comprehensibility (Item 7). Higher scores indicate greater levels of illness perception
Cortisol levels | baseline
  Cortisol is a hormone that is mainly released at times of stress
Cytokine levels of IL-6 and TNF-a | baseline
  Cytokines are a broad and loose category of small proteins (~5-20 kDa) important in cell signaling. Cytokines have been related with anxiety and depression symptoms
Estradiol levels | baseline
  Sexual hormones as estradiol play an important role in mammary carcino- genesis, being able to induce carcinogenic initiation, promotion and progression
Monoamines levels | baseline
  Monoamines refer to the particular neurotransmitters dopamine, noradrenaline and serotonin. These neurotransmitters are involved in different psychopathologies.
Psychological distress scale HADS | four months after
  Hospital Anxiety and Depression Scale ( HADS) was originally developed by Zigmond and Snaith (1983) and is commonly used by doctors to determine the levels of anxiety and depression that a person is experiencing. The total score is out of 42, (21 per anxiety and 21 per depression). Higher scores indicate greater levels of anxiety or depression. Zigmond and Snaith (1983) and is commonly used by doctors to determine the levels of anxiety and depression that a person is experiencing.
Social support perception scale MOS-SSS | four months after
  The Social Support Scale (MOS-SSS) aims to assess the extent to which the person has the support of others to face stressful situations. 19 items with answer categories that range on a 7-point rating scale. Higher scores indicate greater levels of social support perception
Coping scale COPE28 | four months after
  The COPE inventory was created by Carver (1989). It is a multi-dimensional inventory developed to asses the different coping strategies people use in response to stress. Self-distraction, items 1 and 19 Active coping, items 2 and 7 Denial, items 3 and 8 Substance use, items 4 and 11 Use of emotional support, items 5 and 15 Use of instrumental support, items 10 and 23 Behavioral disengagement, items 6 and 16 Venting, items 9 and 21 Positive reframing, items 12 and 17 Planning, items 14 and 25 Humor, items 18 and 28 Acceptance, items 20 and 24 Religion, items 22 and 27 Self-blame, items 13 and 26. Range: 2-8. Higher scores indicate greater levels of coping
Resilience scale | four months after
  The Resilience Scale (RS) was developed to evaluate the levels of resilience in the general population. The items are rated on a 7-point scale ranging 1 (strongly disagree) to 7 (strongly agree), with a score ranging 14 to 98. Higher scores indicate greater levels of resilience
Quality of life scale SF-12 | four months after
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It consists of physical and mental component scores (PCS/MCS), ranging from 0 to 100. Higher scores indicate greater quality of life.
emotional inteligence scale TMMS | four months after
  The Trait Meta-Mood Scale (TMMS; Salovey, Mayer, Goldman, Turvey, & Palfai, 1995) is a well-established measure of perceived emotional intelligence, an aspect of emotional intelligence that includes people's beliefs and attitudes about their own emotional experience. The TMMS-24 contains three key dimensions of emotional intelligence with 8 items each: Emotional Attention, Emotional Clarity and Emotional Repair. The score ranges from 7 to 56. Higher values indicate higher emotional intelligence
illness perception scale | four months after
  The Illness Perception Questionnaire (IPQ) is a widely used multifactorial pencil-and-paper questionnaire which assesses the five cognitive and emotional illness representations and comprehensibility. Five of the items assess cognitive illness representations: consequences (Item 1), timeline (Item 2), personal control (Item 3), treatment control (Item 4), and identity (Item 5). Two of the items assess emotional representations: concern (Item 6) and emotions (Item 8). One item assesses illness comprehensibility (Item 7). Higher scores indicate greater levels of illness perception
Cortisol levels | four months after
  Cortisol is a hormone that is mainly released at times of stress
Cytokine levels of IL-6 and TNF-a | four months after
  Cytokines are a broad and loose category of small proteins (~5-20 kDa) important in cell signaling. Cytokines have been related with anxiety and depression symptoms
Estradiol levels | four months after
  Sexual hormones as estradiol play an important role in mammary carcino- genesis, being able to induce carcinogenic initiation, promotion and progression
Monoamines levels | four months after
  Monoamines refer to the particular neurotransmitters dopamine, noradrenaline and serotonin. These neurotransmitters are involved in different psychopathologies.
Psychological distress scale HADS | through treatment completion, an average of eight months
  Hospital Anxiety and Depression Scale ( HADS) was originally developed by Zigmond and Snaith (1983) and is commonly used by doctors to determine the levels of anxiety and depression that a person is experiencing. The total score is out of 42, (21 per anxiety and 21 per depression). Higher scores indicate greater levels of anxiety or depression.
Social support perception scale MOS-SSS | through treatment completion, an average of eight months
  The Social Support Scale (MOS-SSS) aims to assess the extent to which the person has the support of others to face stressful situations. 19 items with answer categories that range on a 7-point rating scale. Higher scores indicate greater levels of social support perception
Coping scale COPE28 | through treatment completion, an average of eight months
  The COPE inventory was created by Carver (1989). It is a multi-dimensional inventory developed to asses the different coping strategies people use in response to stress. Self-distraction, items 1 and 19 Active coping, items 2 and 7 Denial, items 3 and 8 Substance use, items 4 and 11 Use of emotional support, items 5 and 15 Use of instrumental support, items 10 and 23 Behavioral disengagement, items 6 and 16 Venting, items 9 and 21 Positive reframing, items 12 and 17 Planning, items 14 and 25 Humor, items 18 and 28 Acceptance, items 20 and 24 Religion, items 22 and 27 Self-blame, items 13 and 26. Range: 2-8. Higher scores indicate greater levels of coping
Resilience scale | through treatment completion, an average of eight months
  The Resilience Scale (RS) was developed to evaluate the levels of resilience in the general population. The items are rated on a 7-point scale ranging 1 (strongly disagree) to 7 (strongly agree), with a score ranging 14 to 98. Higher scores indicate greater levels of resilience
Quality of life scale SF-12 | through treatment completion, an average of eight months
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It consists of physical and mental component scores (PCS/MCS), ranging from 0 to 100. Higher scores indicate greater quality of life.
emotional inteligence scale TMMS | through treatment completion, an average of eight months
  The Trait Meta-Mood Scale (TMMS; Salovey, Mayer, Goldman, Turvey, & Palfai, 1995) is a well-established measure of perceived emotional intelligence, an aspect of emotional intelligence that includes people's beliefs and attitudes about their own emotional experience. The TMMS-24 contains three key dimensions of emotional intelligence with 8 items each: Emotional Attention, Emotional Clarity and Emotional Repair. The score ranges from 7 to 56. Higher values indicate higher emotional intelligence
illness perception scale | through treatment completion, an average of eight months
  The Illness Perception Questionnaire (IPQ) is a widely used multifactorial pencil-and-paper questionnaire which assesses the five cognitive and emotional illness representations and comprehensibility. Five of the items assess cognitive illness representations: consequences (Item 1), timeline (Item 2), personal control (Item 3), treatment control (Item 4), and identity (Item 5). Two of the items assess emotional representations: concern (Item 6) and emotions (Item 8). One item assesses illness comprehensibility (Item 7). Higher scores indicate greater levels of illness perception
Cortisol levels | through treatment completion, an average of eight months
  Cortisol is a hormone that is mainly released at times of stress
Cytokine levels of IL-6 and TNF-a | through treatment completion, an average of eight months
  Cytokines are a broad and loose category of small proteins (~5-20 kDa) important in cell signaling. Cytokines have been related with anxiety and depression symptoms
Estradiol levels | through treatment completion, an average of eight months
  Sexual hormones as estradiol play an important role in mammary carcino- genesis, being able to induce carcinogenic initiation, promotion and progression
Monoamines levels | through treatment completion, an average of eight months
  Monoamines refer to the particular neurotransmitters dopamine, noradrenaline and serotonin. These neurotransmitters are involved in different psychopathologies.
Psychological distress scale HADS | four months after treatment completion
  Hospital Anxiety and Depression Scale ( HADS) was originally developed by Zigmond and Snaith (1983) and is commonly used by doctors to determine the levels of anxiety and depression that a person is experiencing. The total score is out of 42, (21 per anxiety and 21 per depression). Higher scores indicate greater levels of anxiety or depression.
Social support perception scale MOS-SSS | four months after treatment completion
  The Social Support Scale (MOS-SSS) aims to assess the extent to which the person has the support of others to face stressful situations. 19 items with answer categories that range on a 7-point rating scale. Higher scores indicate greater levels of social support perception
Coping scale COPE28 | four months after treatment completion
  The COPE inventory was created by Carver (1989). It is a multi-dimensional inventory developed to asses the different coping strategies people use in response to stress. Self-distraction, items 1 and 19 Active coping, items 2 and 7 Denial, items 3 and 8 Substance use, items 4 and 11 Use of emotional support, items 5 and 15 Use of instrumental support, items 10 and 23 Behavioral disengagement, items 6 and 16 Venting, items 9 and 21 Positive reframing, items 12 and 17 Planning, items 14 and 25 Humor, items 18 and 28 Acceptance, items 20 and 24 Religion, items 22 and 27 Self-blame, items 13 and 26. Range: 2-8. Higher scores indicate greater levels of coping
Resilience scale | four months after treatment completion
  The Resilience Scale (RS) was developed to evaluate the levels of resilience in the general population. The items are rated on a 7-point scale ranging 1 (strongly disagree) to 7 (strongly agree), with a score ranging 14 to 98. Higher scores indicate greater levels of resilience
Quality of life scale SF-12 | four months after treatment completion
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It consists of physical and mental component scores (PCS/MCS), ranging from 0 to 100. Higher scores indicate greater quality of life.
emotional inteligence scale TMMS | four months after treatment completion
  The Trait Meta-Mood Scale (TMMS; Salovey, Mayer, Goldman, Turvey, & Palfai, 1995) is a well-established measure of perceived emotional intelligence, an aspect of emotional intelligence that includes people's beliefs and attitudes about their own emotional experience. The TMMS-24 contains three key dimensions of emotional intelligence with 8 items each: Emotional Attention, Emotional Clarity and Emotional Repair. The score ranges from 7 to 56. Higher values indicate higher emotional intelligence
illness perception scale | four months after treatment completion
  The Illness Perception Questionnaire (IPQ) is a widely used multifactorial pencil-and-paper questionnaire which assesses the five cognitive and emotional illness representations and comprehensibility. Five of the items assess cognitive illness representations: consequences (Item 1), timeline (Item 2), personal control (Item 3), treatment control (Item 4), and identity (Item 5). Two of the items assess emotional representations: concern (Item 6) and emotions (Item 8). One item assesses illness comprehensibility (Item 7). Higher scores indicate greater levels of illness perception
Cortisol levels | four months after treatment completion
  Cortisol is a hormone that is mainly released at times of stress
Cytokine levels of IL-6 and TNF-a | four months after treatment completion
  Cytokines are a broad and loose category of small proteins (~5-20 kDa) important in cell signaling. Cytokines have been related with anxiety and depression symptoms
Estradiol levels | fofour months after treatment completion
  Sexual hormones as estradiol play an important role in mammary carcino- genesis, being able to induce carcinogenic initiation, promotion and progression
Monoamines levels | four months after treatment completion
  Monoamines refer to the particular neurotransmitters dopamine, noradrenaline and serotonin. These neurotransmitters are involved in different psychopathologies.
Psychological distress scale HADS | one year after treatment completion
  Hospital Anxiety and Depression Scale ( HADS) was originally developed by Zigmond and Snaith (1983) and is commonly used by doctors to determine the levels of anxiety and depression that a person is experiencing. The total score is out of 42, (21 per anxiety and 21 per depression). Higher scores indicate greater levels of anxiety or depression.
Social support perception scale MOS-SSS | one year after treatment completion
  The Social Support Scale (MOS-SSS) aims to assess the extent to which the person has the support of others to face stressful situations. 19 items with answer categories that range on a 7-point rating scale. Higher scores indicate greater levels of social support perception
Coping scale COPE28 | one year after treatment completion
  The COPE inventory was created by Carver (1989). It is a multi-dimensional inventory developed to asses the different coping strategies people use in response to stress. Self-distraction, items 1 and 19 Active coping, items 2 and 7 Denial, items 3 and 8 Substance use, items 4 and 11 Use of emotional support, items 5 and 15 Use of instrumental support, items 10 and 23 Behavioral disengagement, items 6 and 16 Venting, items 9 and 21 Positive reframing, items 12 and 17 Planning, items 14 and 25 Humor, items 18 and 28 Acceptance, items 20 and 24 Religion, items 22 and 27 Self-blame, items 13 and 26. Range: 2-8. Higher scores indicate greater levels of coping
Resilience scale | one year after treatment completion
  The Resilience Scale (RS) was developed to evaluate the levels of resilience in the general population. The items are rated on a 7-point scale ranging 1 (strongly disagree) to 7 (strongly agree), with a score ranging 14 to 98. Higher scores indicate greater levels of resilience
Quality of life scale SF-12 | one year after treatment completion
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It consists of physical and mental component scores (PCS/MCS), ranging from 0 to 100. Higher scores indicate greater quality of life.
emotional inteligence scale TMMS | one year after treatment completion
  The Trait Meta-Mood Scale (TMMS; Salovey, Mayer, Goldman, Turvey, & Palfai, 1995) is a well-established measure of perceived emotional intelligence, an aspect of emotional intelligence that includes people's beliefs and attitudes about their own emotional experience. The TMMS-24 contains three key dimensions of emotional intelligence with 8 items each: Emotional Attention, Emotional Clarity and Emotional Repair. The score ranges from 7 to 56. Higher values indicate higher emotional intelligence
illness perception scale | one year after treatment completion
  The Illness Perception Questionnaire (IPQ) is a widely used multifactorial pencil-and-paper questionnaire which assesses the five cognitive and emotional illness representations and comprehensibility. Five of the items assess cognitive illness representations: consequences (Item 1), timeline (Item 2), personal control (Item 3), treatment control (Item 4), and identity (Item 5). Two of the items assess emotional representations: concern (Item 6) and emotions (Item 8). One item assesses illness comprehensibility (Item 7). Higher scores indicate greater levels of illness perception
Cortisol levels | one year after treatment completion
  Cortisol is a hormone that is mainly released at times of stress
Cytokine levels of IL-6 and TNF-a | one year after treatment completion
  Cytokines are a broad and loose category of small proteins (~5-20 kDa) important in cell signaling. Cytokines have been related with anxiety and depression symptoms
Estradiol levels | one year after treatment completion
  Sexual hormones as estradiol play an important role in mammary carcino- genesis, being able to induce carcinogenic initiation, promotion and progression
Monoamines levels | one year after treatment completion
  Monoamines refer to the particular neurotransmitters dopamine, noradrenaline and serotonin. These neurotransmitters are involved in different psychopathologies.

CONTACTS AND LOCATIONS:
Locations (1):
- Onkologikoa, San Sebastián, Guipuzcoa, Spain

REFERENCES:
- [Derived] Aizpurua-Perez I, Arregi A, Gonzalez D, Urruticoechea A, Labaka A, Minguez-Alcaide X, Ugartemendia G, Pascual-Sagastizabal E, Echeverria R, Perez-Tejada J. A randomized controlled trial of the effectiveness of a one-to-one peer support intervention on resilience, social support, and salivary cortisol in recently diagnosed women with breast cancer. Eur J Oncol Nurs. 2024 Aug;71:102616. doi: 10.1016/j.ejon.2024.102616. Epub 2024 May 21. PMID 38885598

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT05077371/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT05077371/ICF_001.pdf